CLINICAL TRIAL: NCT00463268
Title: Prevention of Postmenopausal Bone Loss in Osteopenic Women With Alendronate Given on a 70 mg Once-every Two Week Regimen: a 2-year, Double-blind, Placebo-controlled Clinical Trial.
Brief Title: Osteoporosis Prevention With Low Dose Alendronate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Boutsen Yves, professeur, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MG/OP 001
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Osteopenia
Keywords: osteopenia; osteoporosis prevention; alendronate
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Alendronate; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Alendronate 70 mg every 2 weeks
  Interventions: Drug: alendronate; Dietary Supplement: Calcium/Vitamin D
- 2 (Placebo Comparator): Alendronate 70 mg placebo tablet every 2 weeks
  Interventions: Dietary Supplement: Calcium/Vitamin D; Drug: placebo

INTERVENTIONS:
Drug: alendronate — alendronate 70 mg every 2 weeks
  Arms: 1
Dietary Supplement: Calcium/Vitamin D — Calcium 500 mg and vitamin D supplementation according to serum level
Drug: placebo — identical placebo every 2 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of the intermittent administration of alendronate in a low dose, 70 mg once every two week, as osteoporosis prevention for menopausal, osteopenic patients, who don't want or can't receive an oestrogenic substitution treatment.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 60 year-old women
* Menopausal since at least 6 months
* Baseline lumbar BMD from -1 till -2.5

Exclusion Criteria:

* Bone disease other than osteopenia
* Treatment with selective estrogen receptor modulator (SERMs), calcitonin or hormone replacement therapy within 6 monts prior to randomization
* Former or current treatment with any bisphosphonate or bone forming agents
* Chronic use of oral or iv corticosteroids
* Any diagnosis of malignancy less than 12 months

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
percentage of lumbar BMD modification after 2 years | 2 years

SECONDARY OUTCOMES:
percentage of hip BMD modification (total hip and sub-regions) | 2 years
percentage of modification of bone remodeling markers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yves R Boutsen, MD, Principal Investigator
Locations (1):
- University (UCL) Louvain Hospital in Mont-Godinne, Yvoir, Namur, Belgium